CLINICAL TRIAL: NCT06210035
Title: Effects of Heart Rate Oscillations During Meditation on Plasma Biomarkers of Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Mara Mather, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UP-23-00373
Record Dates: First submitted 2023-10-20; First posted 2024-01-18 (Actual); Results first posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Belly-focus concentration meditation (Experimental): Participants will engage in concentration meditation for 40 minutes every day for a week while recording heart rate. They will focus on the sensations around the belly.
  Interventions: Behavioral: Belly-focus meditation
- Belly-focus concentration meditation with slow breathing (Experimental): Participants will engage in concentration meditation and slow breathing for 40 minutes every day for a week while recording heart rate. They will focus on the sensations around the belly while breathing slowly.
  Interventions: Behavioral: Belly-focus meditation with slow breathing
- No-intervention control (No Intervention): Participants will rest quietly for 40 minutes every day for a week while recording heart rate.

INTERVENTIONS:
Behavioral: Belly-focus meditation — Participants will engage in concentration meditation for 40 minutes every day for a week. They will focus on the sensations around the belly.
  Arms: Belly-focus concentration meditation
Behavioral: Belly-focus meditation with slow breathing — Participants will engage in concentration meditation and slow breathing for 40 minutes every day for a week. They will focus on the sensations around the belly while breathing slowly.
  Arms: Belly-focus concentration meditation with slow breathing

SUMMARY:
In the current study, we will examine how two types of concentration meditation practices affect plasma biomarkers of Alzheimer's Disease (AD). We will also examine the effects of the two types of meditation practices on emotional well-being and episodic memory. Healthy adults aged 18-35 who meet all eligibility criteria will be invited to this study. Participants will be asked to engage in one week of daily meditation practice or no-intervention control task at home. They will also be asked to visit the lab twice, once before and once after the intervention, to provide blood samples to assess plasma biomarkers of AD and to complete emotion questionnaires and a memory test.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Aged between 18-35 years old
* Agree to provide blood samples
* Healthy adults who weigh at least 110 pounds
* Agree to devote 40 minutes daily to this study for a week

Exclusion Criteria:

* Have a disorder that would affect heart rhythm or function (e.g., abnormal cardiac rhythm, dyspnea, heart disease including coronary artery disease, angina and arrhythmia)
* Regularly practicing any relaxation, meditation or yoga that involve breathing focused practices lasting for more than an hour each week

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Southern California, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of the 94 participants enrolled, 2 dropped before condition assignment.
Period: Overall Study
Arm/Group | Belly-focus Concentration Meditation | Belly-focus Concentration Meditation With Slow Breathing | No-intervention Control
Started | 30 | 32 | 30
Completed | 27 | 32 | 30
Not Completed | 3 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belly-focus Concentration Meditation | Belly-focus Concentration Meditation With Slow Breathing | No-intervention Control | Total
Number analyzed (Participants) | 30 | 32 | 30 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 32 | 30 | 92
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.07 (5.16) | 26.25 (5.29) | 26.20 (4.82) | 25.73 (5.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 25 | 75
  Male | 6 | 6 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 13 | 8 | 24
  Not Hispanic or Latino | 25 | 18 | 22 | 65
  Unknown or Not Reported | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 13 | 9 | 10 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 0 | 9
  White | 9 | 8 | 10 | 27
  More than one race | 2 | 3 | 4 | 9
  Unknown or Not Reported | 0 | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 30 | 32 | 30 | 92

OUTCOME MEASURES:

1. Primary Outcome: Change in Plasma Amyloid Beta (Aβ) Levels
Description: The investigators computed an aggregate Z-score based on plasma Aβ40 and Aβ42 levels (pg/mL). A Z-score of 0 represents the sample mean. Higher values indicate a greater level of plasma Aβ, which in cognitively normal individuals has been found to be associated with a higher risk of converting to Alzheimer's disease (Song et al., 2011). They conducted a 2 (time: pre, post) × 3 (condition) ANOVA to test for a time × condition interaction in plasma Aβ levels, assessing group differences in change over time.
Time Frame: Measured from blood draws before and after a one-week intervention
Population: Population analyzed is composed by all randomization subjects who completed pre- and post-intervention blood draw and whose data quality was sufficient for data analysis.
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Belly-focus concentration meditation | Belly-focus concentration meditation with slow breathing | No-intervention control
Number analyzed (Participants) | 24 | 28 | 26
Z-score
  pre | -0.38 (0.19) | 0.02 (0.17) | 0.24 (0.18)
  post | -0.08 (0.17) | -0.29 (0.16) | 0.22 (0.16)
Statistical Analysis 1: Comparison: Belly-focus concentration meditation vs Belly-focus concentration meditation with slow breathing vs No-intervention control; Test type: Superiority; p = 0.003, ANOVA; F test = 6.21

2. Primary Outcome: Change in Plasma Ab42/40 Ratio
Description: The investigators conducted a 2 (time: pre, post) × 3 (condition) ANOVA to test for an interaction effect on plasma Ab42/40 ratios. The plasma Ab42/40 ratio was calculated by dividing the plasma Ab42 concentration (pg/ml) by the plasma Ab40 concentration (pg/ml). A higher plasma Ab42/40 ratio indicates better outcome (i.e., greater brain clearance).
Time Frame: Measured from blood draws before and after a one-week intervention
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ratio of Aβ42 to Aβ40
Arm/Group | Belly-focus concentration meditation | Belly-focus concentration meditation with slow breathing | No-intervention control
Number analyzed (Participants) | 22 | 28 | 25
ratio of Aβ42 to Aβ40
  pre | 0.05 (0.002) | 0.05 (0.001) | 0.05 (0.001)
  post | 0.05 (0.002) | 0.05 (0.001) | 0.05 (0.002)
Statistical Analysis 1: Comparison: Belly-focus concentration meditation vs Belly-focus concentration meditation with slow breathing vs No-intervention control; Test type: Superiority; p = 0.460, ANOVA; F test = 0.78

3. Secondary Outcome: Change in Plasma pTau-181/Tau Ratio
Description: The investigators conducted a 2 (time: pre, post) × 3 (condition) ANOVA to test for an interaction effect on plasma pTau-181/total Tau ratios. The plasma pTau-181/total Tau ratio was calculated by dividing the plasma pTau-181 concentration (pg/ml) by the plasma total Tau concentration (pg/ml). A higher plasma pTau-181/total Tau ratio indicates better outcome (i.e., greater brain clearance).
Time Frame: Measured from blood draws before and after a one-week intervention
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ratio of pTau-181 to total Tau
Arm/Group | Belly-focus concentration meditation | Belly-focus concentration meditation with slow breathing | No-intervention control
Number analyzed (Participants) | 23 | 25 | 23
ratio of pTau-181 to total Tau
  pre | 5.30 (0.38) | 4.78 (0.37) | 5.02 (0.38)
  post | 4.73 (0.37) | 5.29 (0.36) | 4.64 (0.37)
Statistical Analysis 1: Comparison: Belly-focus concentration meditation vs Belly-focus concentration meditation with slow breathing vs No-intervention control; Test type: Superiority; p = 0.127, ANOVA; F test = 2.13

4. Secondary Outcome: Change in Emotional Well-being
Description: The investigators conducted a 2 (time: pre, post) × 3 (condition) ANOVA to test for an interaction effect on emotional well-being. Emotional well-being was assessed using the Profile of Mood States (POMS), which consists of 40 items rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Total Mood Disturbance (TMD) scores were calculated by summing the negative mood items and subtracting the sum of the positive mood items. A constant of 100 was added to the TMD score to eliminate negative values. Higher scores indicate more negative mood states, with possible scores ranging from 56 to 216.
Time Frame: Measured before and after a one-week intervention
Population: Population analyzed is composed by all randomization subjects who completed the emotional well-being survey (i.e., POMS) at pre- and post-intervention and whose data quality was sufficient for data analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Belly-focus concentration meditation | Belly-focus concentration meditation with slow breathing | No-intervention control
Number analyzed (Participants) | 27 | 31 | 26
score on a scale
  pre | 87.15 (2.29) | 87.39 (2.14) | 94.73 (2.34)
  post | 89.89 (2.93) | 84.68 (2.73) | 94.96 (2.99)
Statistical Analysis 1: Comparison: Belly-focus concentration meditation vs Belly-focus concentration meditation with slow breathing vs No-intervention control; Test type: Superiority; p = 0.952, ANOVA; F test = 0.004

5. Other Pre Specified Outcome: Episodic Memory
Description: The investigators will conduct a one-way ANOVA to assess group differences in episodic memory.
Time Frame: Measured after a one-week intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: One week
Arm/Group | Belly-focus Concentration Meditation | Belly-focus Concentration Meditation With Slow Breathing | No-intervention Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/32 | 0/30
Other Adverse Events (participants affected / at risk) | 3/30 | 0/32 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belly-focus Concentration Meditation (N=30) | Belly-focus Concentration Meditation With Slow Breathing (N=32) | No-intervention Control (N=30)
Adverse events after blood draw (Blood and lymphatic system disorders) | 3 | 0 | 0 — Three participants reported mild events after blood draws: two had brief discomfort or bleeding; one fainted briefly, recovered after snacks, and was cleared by paramedics. All recovered fully; no serious adverse events occurred.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT06210035/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT06210035/SAP_001.pdf